CLINICAL TRIAL: NCT03460301
Title: Observational of GPI-anchored Protein-deficient (PNH-Type) Cells in Korean Patients With Bone Marrow Failure Syndrome and Having Hemolytic Paroxymal Nocturnal Hemoglobinuria (OPENK)
Brief Title: Observational of PNH Type Cells in Korean Patients With Bone Marrow Failure Syndrome and Having Hemolytic PNH
Acronym: OPENK
Status: Completed | Type: Observational
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OPENK
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: PNH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who are positive of PNH-type cells are followed up for the percentage of PNH-type cells regularly for examining how it change.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Commbs' test - negative
* Any patients meeting any of Idiopathic AA/MDS/Patients who had PNH clone size <10%

Exclusion Criteria:

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Idiopatic AA/MDS/Patients who had PNH clone size <10%
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Time-course changes in the percentage of PNH-type cells in patients who are positive of PNH-type cells during period | 5 years

IPD SHARING:
Plan to Share IPD: No